CLINICAL TRIAL: NCT06131411
Title: Cardio-metabolic Diseases in Immigrants and Ethnic Minorities: From Epidemiology to New Prevention Strategies
Acronym: DIABETHIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Collaborators: Azienda Ospedaliera Universitaria Renato Dulbecco (Unknown); AUSL - IRCCS in Tecnologie Avanzate e Modelli Assistenziali in Oncologia di Reggio Emilia (Unknown); Istituto Nazionale per la promozione della salute delle popolazioni Migranti e per il contrasto delle malattie della Povertà (INMP) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: DIABETHIC
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: health promotion; ethnic minorities; cardiovascular diseases; obesity; hypertension; Migrant health; Ambulatory care-sensitive conditions; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Obesity; Hypertension; Ambulatory Care Sensitive Conditions | interventions — Health Promotion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Health promotion intervention
  Interventions: Other: Health promotion
- Control (Placebo Comparator): Usual care
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Health promotion — Co-created culture-tailored intervention of health promotion aimed to increase healthy diet, physical activity and compliance with treatment protocols for diabetes.
  Arms: Intervention
Other: Usual care — Health promotion activities routinely performed by Diabetes clinics at the recruiting centres.
  Arms: Control

SUMMARY:
The purpose of this clinical trial is to learn if intervention on health behavior can promote diabetes care and improve compliance to therapeutic protocols in ethnic minorities with type 2 diabetes. To answer this question, researchers will compare the effectiveness of co-created, culture-sensitive intervention to that of a usual-care approach to promote diabetes care 12 months after enrollment in first-generation immigrants with type 2 diabetes.

DETAILED DESCRIPTION:
Diabetes mellitus has an unequal impact globally, with 80% of cases occurring in low- and middle-income countries. In particular, social determinants of health, such as education, employment, and living conditions, play a significant role in the unequal impact of diabetes. On the other hand, cultural aspects such as education on healthy behaviors, diet, adherence to drug therapy, self-monitoring of blood glucose, and physical activity, are essential for effective diabetes management. Finally, beliefs about the disease, communication difficulties, limited educational backgrounds, and the inability to understand educational materials and read food labels due to language barriers can pose obstacles to achieving adequate disease awareness and control among ethnic minorities. Large randomized clinical trials conducted over the past decade have examined the effectiveness of behavioral interventions to address these influences among diverse ethnic minorities. These studies, mainly conducted on specific ethnic groups living in the US such as Afro-American and Hispanic populations, reported improvements in glycosylated hemoglobin A1c control at 3- and at 6-months post intervention compared with control groups who received 'usual care', being sustained to a lesser extent at 12- and 24-months post intervention. In Europe, where diabetes disproportionately affects adult populations from ethnic minorities, with higher disease risk and complication and mortality rates compared to European host populations, studies on culturally sensitive diabetes self-management education and support are limited, and their effectiveness remains uncertain. The multicenter randomized clinical trial (DiabEthic trial) was therefore designed to compare the effectiveness of culture-sensitive intervention to that of a usual-care approach to promote diabetes care and to improve compliance to therapeutic protocols in first-generation immigrants with type 2 diabetes. To best transfer this experience into clinical practice, personalized cultural approaches to type 2 diabetes were developed with the support of representatives of ethnic communities living in Italy and the participation of specific cultural mediators. Unlike previous studies, this multicenter study focuses on the diversely represented ethnic communities in different parts of Italy.

ELIGIBILITY:
Inclusion Criteria:

* Immigrant status: Self-identification of being born in High migration pressure countries from parents born in high migration pressure countries
* Age ≥ 18 years
* Type 2 diabetes newly diagnosed or with HbA1c > 8% in the last assessment within 24 months before the visit

Exclusion Criteria:

* Patients who will not provide the informed consent
* Patients with HbA1c ≤ 8% in the last assessment within 24 months before the visit
* Severe psychiatric disorders
* Pregnant women
* Critical illness
* Impaired cognitive or physical ability that could make the intervention not feasible, as judged by clinical staff members

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Glycated haemoglobin (HbA1c) | from baseline to follow-up at month 12
  Change in glycated haemoglobin (HbA1c)

SECONDARY OUTCOMES:
Systolic Blood Pressure | from baseline to follow-up at month 12
  Change in Systolic Blood Pressure
Diastolic Blood Pressure | from baseline to follow-up at month 12
  Change in Diastolic Blood Pressure
Total Cholesterol | from baseline to follow-up at month 12
  Change in Total Cholesterol
LDL Cholesterol | from baseline to follow-up at month 12
  Change in LDL Cholesterol
HDL Cholesterol | from baseline to follow-up at month 12
  Change in HDL Cholesterol
Triglycerides | from baseline to follow-up at month 12
  Change in triglycerides
Body Mass Index (BMI) | from baseline to follow-up at month 12
  Change in Body Mass Index (BMI)
Waist circumference | from baseline to follow-up at month 12
  Change in Waist circumference
Physical activity | from baseline to follow-up at month 12
  Change in compliance with World Health Organization recommended exercise goals
Adherence to Mediterranean Diet | from baseline to follow-up at month 12
  Change in Adherence to Mediterranean Diet

CONTACTS AND LOCATIONS:
Overall Officials: Pietro A Modesti, MD, PhD, Principal Investigator — Azienda Ospedaliero-Universitaria Careggi
Locations (4):
- Italy (4):
  - Azienda Ospedaliera Universitaria Renato Dulbecco, Catanzaro, Catanzaro
  - Azienda Ospedaliera-Universitaria Careggi, Florence, Florence
  - AUSL - IRCCS in Tecnologie Avanzate e Modelli Assistenziali in Oncologia di Reggio Emilia, Reggio Emilia, Reggio Emilia
  - Istituto Nazionale per la promozione della salute delle popolazioni Migranti e il contrasto delle malattie della Povertà (INMP), Rome, Rome

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bonvicini L, Venturelli F, Bononi F, Balestra GL, Iorio G, Ghirotto L, Petrelli A, Pierconti S, Laurendi G, Perticone M, Pellegrino A, Boddi M, Modesti PA, Giorgi Rossi P; DIABETHIC Working Group. A randomized trial to evaluate a complex, co-created, culture-sensitive intervention to promote healthy lifestyles and compliance to therapy in immigrants with type 2 diabetes: A protocol of a multicenter Italian study. PLoS One. 2025 Feb 24;20(2):e0317994. doi: 10.1371/journal.pone.0317994. eCollection 2025. PMID 39992940